CLINICAL TRIAL: NCT03062215
Title: Assessing the Efficacy of a Culturally Adapted Cognitive Behavioural Internet-delivered Treatment for Depression: Protocol for a Randomised Controlled Trial
Brief Title: Efficacy of a Culturally Adapted Cognitive Behavioural Internet-delivered Treatment for Depression
Acronym: CAiCBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silver Cloud Health (Other)
Collaborators: Irish Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAiCBT
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Depression
Keywords: Culturally adapted psychotherapy; Internet-delivered treatment; Depression; Latin America
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Space from depression (Experimental): SilverCloud Health is a leading provider of online therapeutic solutions to support and promote positive behavior change and mental wellness. SilverCloud delivers interventions depression. The treatment includes self-monitoring, behavioural activation, cognitive restructuring, and challenging core beliefs. All modules have the same structure and format, which consist of quizzes, videos, educational content, activities with homework suggestions and a module review page. Also, users have a supporter, who will give feedback asynchronously (D Richards et al., 2015). Research on the SilverCloud interventions has yielded significant clinical outcomes (D Richards et al., 2015).
  Interventions: Behavioral: Space from Depression
- Control Group (No Intervention): Waiting list

INTERVENTIONS:
Behavioral: Space from Depression — Space from Depression programme (Yo puedo sentirme Bien -Spanish version) consists of seven modules of cognitive-behavioural therapy. The treatment includes self-monitoring, behavioural activation, cognitive restructuring, and challenging core beliefs. All modules have the same structure and format, which consist of quizzes, videos, educational content, activities with homework suggestions and a module review page.
  Other Names: Yo puedo sentirme bien
  Arms: Space from depression

SUMMARY:
The study seeks to evaluate the efficacy of a culturally adapted internet-delivered treatment for depression in Colombia. The research involves two studies: (a) the cultural adaptation of the Space from Depression cognitive-behavioural internet-delivered programme, and (b) the implementation of the culturally adapted intervention using a randomised controlled trial methodology. The study will be a first contribution of a culturally adapted low-intensity internet-delivered intervention with Latin Americans.

DETAILED DESCRIPTION:
Depression is the principal cause of disability in the world. High rates of prevalence of depression in general populations and college students have been found worldwide and in various cultural groups. For instance, a 12-month prevalence rate has been estimated in the U.S. at 9.5% and in Europe at 8.5% of the population. In Colombia, 12-month prevalence is between 6.2% and 12.1%. The Colombian National Mental Health Survey has estimated point prevalence of mild to moderate depressive symptoms at 15.6% and severe depressive symptoms at 4.2% of adults. On the other hand, there are significant barriers for accessing mental health services in Colombia. About 50% of the population does not have access to health services, while the majority of the population with mental health problems do not have adequate mental health insurance coverage.

Although low-intensity interventions for depression have been developed in western high-income countries and these interventions therefore have been influenced by their specific cultural context (for example, Ireland, UK, Australia), it is important to consider how cultural context may impact on the adaptation for use in LMICs such as Colombia. The authors argue that cultural aspects need to be taken into consideration when translating and adapting interventions to help guarantee similar results to what have been achieved in high-income countries.

General method Aims and Hypothesis: We aim to assess the efficacy of a culturally adapted cognitive behavioural internet-delivered treatment for college students with depressive symptoms in Colombia. In line with other studies in high-income countries (HICs), and using an already established intervention, we hypothesise that the culturally adapted Space from Depression programme will be efficacious, with significant changes within the treatment group and differences post-treatment between the active treatment and the waiting list control group.

The study is a mixed method approach utilising in study 1, quantitative and qualitative methods to assist in the cultural adaptation of the Space from Depression intervention and in study 2 a randomised control design to examine the efficacy of the culturally-adapted intervention.

Procedure The programme Space from Depression will be culturally adapted for a Colombian population using cultural sensitivity and ecological validity frameworks, including principles from cross-cultural assessment research. (Study 1). Once the programme is culturally adapted, it will be tested using a randomised controlled trial methodology (Study 2).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above
* Mild to moderately severe depressive symptoms: (PHQ-9 score 10-19)

Exclusion Criteria:

* Severe depressive symptoms >19 on PHQ-9
* Suicidal ideation or intent: Score of 2 or above on PHQ-9 question 9
* Psychosis
* Currently in psychological treatment for depression
* On medication for less than 1 month
* Alcohol or drugs misuse
* Previous diagnosis of an organic mental health disorder
* Depression preceding or coinciding a diagnosed medical condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire -9 | 6 months
  depression symptoms

SECONDARY OUTCOMES:
Generalised Anxiety Disorder 7 | 6 months
  anxiety symptoms

OTHER OUTCOMES:
Satisfaction with Treatment Questionnaire | 2 months
  Patient satisfaction
Helpful Aspects of Therapy Questionnaire | weekly for 7 weeks
  Significant events

CONTACTS AND LOCATIONS:
Overall Officials: Derek Richards, PhD, Study Director — University of Dublin, Trinity College; Alicia Salamanca, MSc, Principal Investigator — University of Dublin, Trinity College
Locations (2):
- Colombia (2):
  - University Los Andes, Bogotá
  - University of Bucaramanga, Bucaramanga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayuso-Mateos JL, Vazquez-Barquero JL, Dowrick C, Lehtinen V, Dalgard OS, Casey P, Wilkinson C, Lasa L, Page H, Dunn G, Wilkinson G; ODIN Group. Depressive disorders in Europe: prevalence figures from the ODIN study. Br J Psychiatry. 2001 Oct;179:308-16. doi: 10.1192/bjp.179.4.308. PMID 11581110
- [Background] Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):617-27. doi: 10.1001/archpsyc.62.6.617. PMID 15939839
- [Background] Bromet E, Andrade LH, Hwang I, Sampson NA, Alonso J, de Girolamo G, de Graaf R, Demyttenaere K, Hu C, Iwata N, Karam AN, Kaur J, Kostyuchenko S, Lepine JP, Levinson D, Matschinger H, Mora ME, Browne MO, Posada-Villa J, Viana MC, Williams DR, Kessler RC. Cross-national epidemiology of DSM-IV major depressive episode. BMC Med. 2011 Jul 26;9:90. doi: 10.1186/1741-7015-9-90. PMID 21791035
- [Background] Demyttenaere K, Bruffaerts R, Posada-Villa J, Gasquet I, Kovess V, Lepine JP, Angermeyer MC, Bernert S, de Girolamo G, Morosini P, Polidori G, Kikkawa T, Kawakami N, Ono Y, Takeshima T, Uda H, Karam EG, Fayyad JA, Karam AN, Mneimneh ZN, Medina-Mora ME, Borges G, Lara C, de Graaf R, Ormel J, Gureje O, Shen Y, Huang Y, Zhang M, Alonso J, Haro JM, Vilagut G, Bromet EJ, Gluzman S, Webb C, Kessler RC, Merikangas KR, Anthony JC, Von Korff MR, Wang PS, Brugha TS, Aguilar-Gaxiola S, Lee S, Heeringa S, Pennell BE, Zaslavsky AM, Ustun TB, Chatterji S; WHO World Mental Health Survey Consortium. Prevalence, severity, and unmet need for treatment of mental disorders in the World Health Organization World Mental Health Surveys. JAMA. 2004 Jun 2;291(21):2581-90. doi: 10.1001/jama.291.21.2581. PMID 15173149
- [Background] Bernal, Sáez-Santiago E. Culturally centered psychosocial interventions. Journal of Community Psychology. 2006;34(2):121.
- [Background] Richards D, Timulak L, Hevey D. A comparison of two online cognitive-behavioural interventions for symptoms of depression in a student population: The role of therapist responsiveness. Counselling & Psychotherapy Research. 2013;13(3):184-93.
- [Background] Ministry of Health. National Mental Health survey. Bogota, Colombia: Ministry of Health; 2015. Report No.: 978-958-8903-19-4.
- [Background] Rodriguez J. La atención de Salud Mental en América Latina y el caribe. Rev Psiquiatr Urug. 2007;71(2):117-24.
- [Background] Merz EL, Malcarne VL, Roesch SC, Riley N, Sadler GR. A multigroup confirmatory factor analysis of the Patient Health Questionnaire-9 among English- and Spanish-speaking Latinas. Cultur Divers Ethnic Minor Psychol. 2011 Jul;17(3):309-316. doi: 10.1037/a0023883. PMID 21787063
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Gilbody S, Richards D, Brealey S, Hewitt C. Screening for depression in medical settings with the Patient Health Questionnaire (PHQ): a diagnostic meta-analysis. J Gen Intern Med. 2007 Nov;22(11):1596-602. doi: 10.1007/s11606-007-0333-y. Epub 2007 Sep 14. PMID 17874169
- [Background] Richards D, Timulak L, O'Brien E, Hayes C, Vigano N, Sharry J, Doherty G. A randomized controlled trial of an internet-delivered treatment: Its potential as a low-intensity community intervention for adults with symptoms of depression. Behav Res Ther. 2015 Dec;75:20-31. doi: 10.1016/j.brat.2015.10.005. Epub 2015 Oct 21. PMID 26523885
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Garcia-Campayo J, Zamorano E, Ruiz MA, Pardo A, Perez-Paramo M, Lopez-Gomez V, Freire O, Rejas J. Cultural adaptation into Spanish of the generalized anxiety disorder-7 (GAD-7) scale as a screening tool. Health Qual Life Outcomes. 2010 Jan 20;8:8. doi: 10.1186/1477-7525-8-8. PMID 20089179
- [Background] Llewelyn SP. Psychological therapy as viewed by clients and therapists. Br J Clin Psychol. 1988 Sep;27(3):223-37. doi: 10.1111/j.2044-8260.1988.tb00779.x. PMID 3191302
- [Background] Elliott R, Slatick E, Urman M. Qualitative change process research on psychotherapy: Alternative strategies. Psychological Test and Assessment Modeling. 2001;43(3):69.
- [Background] Richards D, Timulak L. Satisfaction with therapist-delivered vs. self-administered online cognitive behavioural treatments for depression symptoms in college students. British Journal of Guidance & Counselling. 2013;41(2):193-207.
- [Derived] Salamanca-Sanabria A, Richards D, Timulak L, Connell S, Mojica Perilla M, Parra-Villa Y, Castro-Camacho L. A Culturally Adapted Cognitive Behavioral Internet-Delivered Intervention for Depressive Symptoms: Randomized Controlled Trial. JMIR Ment Health. 2020 Jan 31;7(1):e13392. doi: 10.2196/13392. PMID 32003749
- [Derived] Salamanca-Sanabria A, Richards D, Timulak L, Castro-Camacho L, Mojica-Perilla M, Parra-Villa Y. Assessing the efficacy of a culturally adapted cognitive behavioural internet-delivered treatment for depression: protocol for a randomised controlled trial. BMC Psychiatry. 2018 Feb 27;18(1):53. doi: 10.1186/s12888-018-1634-x. PMID 29482586